CLINICAL TRIAL: NCT07297355
Title: UVIS - UCLouvain Vertigo International Survey
Brief Title: Four Ways to Be Dizzy: When Physiology Fails to Explain Disability Insights From the UVIS International Survey
Acronym: UVIS
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ABMA-3
Record Dates: First submitted 2025-12-01; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Vestibular Disease; Vestibular Dysfunction
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vestibular: Patients with vestibular loss diagnosed by senior ENT doctors with the gold standard ENT measures (caloric testing, head impulse test and/or vestibular evoked myogenic potential, ocular and cervical)
- Healthy controls: People with no vestibular loss

SUMMARY:
The aim of this international study is to better understand how vestibular disorders affect daily life, including physical balance, vision and movement tolerance, emotional wellbeing, and cognitive functioning. Vestibular disorders are common but often difficult to diagnose because symptoms vary widely from one patient to another. To improve clinical care, we need large-scale information on the real-world experience of patients across different countries and clinical settings.

The UCLouvain Vertigo International Survey (UVIS) collects standardized information from adults with confirmed vestibular disorders, including questionnaires about dizziness-related handicap, emotional symptoms, and cognitive-vestibular complaints. Ear-nose-throat (ENT) specialists also provide routine clinical test results, such as caloric testing, vestibular evoked myogenic potentials (cVEMP and oVEMP), video head impulse tests (vHIT), and posturography. By combining these data, the study aims to identify different patient profiles and to examine how subjective symptoms relate to the physiological function of the vestibular system.

Participants take part during their routine clinical visit. They complete short questionnaires (on dizziness, anxiety, depression, cognitive symptoms, and daily functioning), and their ENT specialist encodes the results of the vestibular tests already performed as part of their usual care. No additional medical tests are required for the study.

By comparing data from several centers in Belgium, France, and the United States, this project seeks to provide a more complete picture of vestibular disorders worldwide and to support the development of better diagnostic tools and more personalized rehabilitation strategies.

ELIGIBILITY:
For patients :

Inclusion Criteria:

* Age between 18 and 90 years old.
* Vestibular loss diagnosed by senior ENT doctors

Exclusion Criteria:

* Previous neurological disorders (stroke, dementia, …)
* Current medication interfering with the testing (reducing reaction time).
* Visual difficulties interfering with the testing (Visual field reduction,…)
* Age below 18 years old.

For healthy controls :

Inclusion criteria :

- Age between 18 and 90 years old.

Exclusion criteria:

* Previous neurological disorders (stroke, dementia, …)
* Current medication interfering with the testing (reducing reaction time)
* Visual difficulties interfering with the testing (Visual field reduction,…)
* Vertigo or balance complains or an history of previous vestibular disorder.
* Age below 18 years old.
* Not being able to understand the consigns of the task.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vestibular loss diagnosed by senior ENT doctors
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-08-03 (Actual); Study Completion 2025-08-03 (Actual)

PRIMARY OUTCOMES:
Assessment of dizziness-related handicap | Through the entire study, approximately 36 months.
  DHI - Dizziness Handicap Inventory (25 items; physical, functional, emotional subscales). Scores 0-100. Higher scores = greater handicap.
Assessment of emotional symptoms | Through the entire study, approximately 36 months.
  HADS - Hospital Anxiety and Depression Scale (14 items; Anxiety and Depression subscales). Scores 0-21 per subscale. Higher scores = more symptoms
Assessment of cognitive-vestibular complaints | Through the entire study, approximately 36 months.
  NVI - Neuropsychological Vertigo Inventory (22 items assessing cognitive-vestibular symptoms: attention, memory, spatial orientation, visuospatial abilities). Higher scores = more complaints

SECONDARY OUTCOMES:
Vestibular Physiological Function - canal paresis percentage | Through the entire study, approximately 36 months.
Vestibular Physiological Function - cVEMP and oVEMP | Through the entire study, approximately 36 months.
Vestibular Physiological Function - video Head Impulse Test | Through the entire study, approximately 36 months.
Vestibular Physiological Function - Posturography | Through the entire study, approximately 36 months.

CONTACTS AND LOCATIONS:
Locations (3):
- Medical University of South Carolina, Charleston, South Carolina, United States
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Hopital européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No